CLINICAL TRIAL: NCT04564898
Title: A Phase I/II Study Exploring the Safety and Activity of Trifluridine/Tipiracil in Combination With Capecitabine and Bevacizumab in Metastatic Colorectal Cancer Patients
Brief Title: Trifluridine/Tipiracil in Combination With Capecitabine and Bevacizumab in Metastatic Colorectal Cancer Patients.
Acronym: TriComB
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-513271-41-00
Record Dates: First submitted 2020-09-12; First posted 2020-09-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Capecitabine; Bevacizumab; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- trifluridine/tipiracil plus capecitabine and bevacizumab (Experimental)
  Interventions: Drug: Capecitabine; Drug: Bevacizumab; Drug: Trifluridine/Tipiracil

INTERVENTIONS:
Drug: Capecitabine — Part 1 • Capecitabine, 1000 mg/sqm orally twice daily on days 1-14 each 28 days
  Part 2
  • Capecitabine, 1000 mg/sqm orally twice daily on days 1-14 each 28 days
Drug: Bevacizumab — Part 1 • Bevacizumab, 5 mg/kg IV dose over 30 minutes on days 1 and 15 each 28 days
  Part 2
  • Bevacizumab, 5 mg/kg IV dose over 30 minutes on days 1 and 15 each 28 days
Drug: Trifluridine/Tipiracil — Part 1 • Trifluridine/tipiracil, dose escalation from 25 mg/sqm to 35 mg/sqm orally twice daily on days 15-19 (and days 22-26) each 28 days
  Part 2
  • Trifluridine/tipiracil, at the recommanded dose established during part 1 orally twice daily on days 15-19 (and days 22-26) each 28 days

SUMMARY:
The aim oh this study is to determine the safety and recommended dose of trifluridine/tipiracil plus capecitabine and bevacizumab combination (part 1, dose escalation phase) and to assess its activity in previously untreated mCRC patients who are deemed not eligible for intensive chemotherapy (part 2, expansion phase).

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase 1/2 study evaluating the safety and activity of trifluridine/tipiracil in combination with capecitabine and bevacizumab in mCRC. The first part (Part 1) of the study will consist in a dose-escalation assessment of the safety of the treatment in subjects with previously untreated mCRC deemed not fit for irinotecan- and/or oxaliplatin- based regimens (i. e. FOLFOX/XELOX/FOLFIRI/FOLFOXIRI with or without targeted agents).

The second part (Part 2) will be an open-label phase 2 study with a Fleming's single-stage design to evaluate the ORR of the study treatment at the recommended dose established in the first part of the study in the same patients' population.

Trifluridine/tipiracil, capecitabine and bevacizumab will be administered in 28-days cycles until progressive disease, unacceptable toxicities, or patients' refusal.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to study procedures.
* Histologically proven diagnosis of colorectal cancer.
* Metastatic colorectal cancer not previously treated with chemotherapy for metastatic disease.
* At least one measurable lesion according to RECIST1.1.
* Age ≥ 18 years.
* ECOG PS ≤ 1.
* Life expectancy of at least 12 weeks.
* Previous adjuvant fluoropyrimidine-based chemotherapy allowed only if more than 12 months elapsed between the end of adjuvant and first relapse.
* Availability of archival tumour tissue (primary tumour and metastases or at least one of the two) for biomarker analysis.
* Availability of blood sample for biomarker analysis.
* Previously not eligible for a chemotherapy doublet or triplet (oxaliplatin and/or irinotecan-based combination).
* Neutrophils ≥1.5 x 109/L, Platelets ≥100 x 109/L, Hemoglobin ≥ 9 g/dl.
* Total bilirubin ≤1.5 fold the upper-normal limits (UNL), AST (SGOT) and/or ALT (SGPT) ≤ 2.5 x UNL (or <5 x UNL in the case of liver metastases), alkaline phosphatase ≤ 2.5 x UNL (or <5 x UNL in case of liver metastases).
* Creatinine clearance ≥ 50 mL/min or serum creatinine ≤1.5 x UNL.
* Male subjects with female partners of childbearing potential must be willing to use adequate contraception as approved by the investigator (barrier contraceptive measure or oral contraception).
* Women of childbearing potential must have a negative blood pregnancy test at the baseline visit. For this trial, women of childbearing potential are defined as all women after puberty, unless they are postmenopausal for at least 12 months, are surgically sterile, or are sexually inactive.
* Subjects and their partners must be willing to avoid pregnancy during the trial and until 6 months after the last trial treatment.
* Will and ability to comply with the protocol.

Exclusion Criteria:

* Radiotherapy to any site within 4 weeks before the study.
* Previous treatment with trifluridine/tipiracil, bevacizumab and capecitabine (previous treatment with capecitabine was permitted only in the adjuvant setting and if more than 12 months elapsed between the end of adjuvant and first relapse).
* Untreated brain metastases or spinal cord compression or primary brain tumors.
* History or evidence upon physical examination of CNS disease unless adequately treated.
* Clinical signs of malnutrition.
* Active uncontrolled infections or other clinically relevant concomitant illness contraindicating chemotherapy administration.
* Evidence of bleeding diathesis or coagulopathy.
* Uncontrolled hypertension and prior history of hypertensive crisis or hypertensive encephalopathy.
* Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication.
* Significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months of study enrolment.
* Any previous venous thromboembolism ≥ NCI CTCAE Grade 4.
* History of abdominal fistula, GI perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to the first study treatment.
* Treatment with any investigational drug within 30 days prior to enrolment or 2 investigational agent half-lives (whichever is longer).
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.
* Known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs.
* Any concomitant drugs contraindicated for use with the trial drugs according to the product information of the pharmaceutical companies.
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Sexually active males and females (of childbearing potential) unwilling to practice contraception (barrier contraceptive measure or oral contraception) during the study and until 6 months after the last trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
recommended dose | 2 years
  recommended dose of the combination trifluridine/tipiracil plus capecitabine plus bevacizumab
activity | 3 years
  activity of the combination trifluridine/tipiracil plus capecitabine plus bevacizumab in terms of overaal response rate per RECIST v1.1.

SECONDARY OUTCOMES:
quality of life for cancer patients | 3 years
  quality of life as measured by EORTC QLQ-C30 questionnaire.
quality of life for colorectal cancer patients | 3 years
  quality of life as measured by EORTC QLQ-CR29 questionnaire.
quality of life for dimensions health | 3 years
  quality of life as measured by EuroQol EQ-5D questionnaire.
survival | 3 years
  efficacy of the combination trifluridine/tipiracil plus capecitabine plus bevacizumab in terms of progression-free survival and overall survival

OTHER OUTCOMES:
bioavailability | 2 years
  Absolute and relative bioavailability of the combination trifluridine/tipiracil plus capecitabine plus bevacizumab.
Steady state concentration | 2 years
  Steady state concentration of the combination trifluridine/tipiracil plus capecitabine plus bevacizumab.
Therapeutic index | 2 years
  Therapeutic index of the combination trifluridine/tipiracil plus capecitabine plus bevacizumab.
Volume of distribution | 2 years
  Volume of distribution of the combination trifluridine/tipiracil plus capecitabine plus bevacizumab.
Half-life | 2 years
  Plasma half-life of the combination trifluridine/tipiracil plus capecitabine plus bevacizumab.
Clearance | 2 years
  Clearance of the combination trifluridine/tipiracil plus capecitabine plus bevacizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Cremolini, MD, PhD, Study Chair — Fondazione GONO
Locations (2):
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan, MI
  - Azienda Ospedaliero Universitaria Pisana, Pisa, PI

IPD SHARING:
Plan to Share IPD: No